CLINICAL TRIAL: NCT02661906
Title: Effect of SKY on Anxiety, Depression and Quality of Life of Type 2 Diabetic Patients After a 6 Days Intervention
Brief Title: A Pilot Study on Effect of SKY on Psychosocial Parameters of Type 2 Diabetic Patients After a 6 Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RA 2014-028
Record Dates: First submitted 2015-10-08; First posted 2016-01-25 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SKY Pre (Experimental): Sudarshan Kriya Yoga is provided to all the enrolled participants. The baseline characteristics of patient is compared with that of their characteristics after yoga intervention. All the participants were provided with yoga training for 6 days and then asked to perform the SKY at home daily till 12 week. The questionnaire on anxiety, depression and quality of life were administered at the baseline and at the end of 6 days of yoga. Biochemical parameters such as HbA1c, lipid profile, fasting glucose and post meal glucose were measured at baseline and after 12 week of intervention.
  Interventions: Other: SKY
- SKY post (Active Comparator): The enrolled participants were provided with SKY intervention and their pre and post data were recorded.
  Interventions: Other: SKY

INTERVENTIONS:
Other: SKY — Sudarshan Kriya Yoga is a rhythmic breathing exercise with slow and fast breath at a particular pace.It is recommended for stress management as yoga is a mind body control tool. SKY is having effect on multiple organ thus causing the positive effect.

SUMMARY:
The purpose of this study is to determine whether Sudarshan Kriya Yoga intervention has effect on the quality of life , anxiety and depression of Type 2 Diabetic Patients.

DETAILED DESCRIPTION:
Diabetes is a psychologically and behaviorally demanding disease; therefore psychosocial factors are relevant to nearly all aspects of its management. Research findings have demonstrated that depression is more common in patients with diabetes than in the general population, at least 15 % of patients have clinical depression.Yoga is a mind-body alternative therapy which can be used to prevent and treat type 2 diabetes mellitus and related complications.

Sudarshan kriya Yoga is a unique yogic breathing practices which involves several types of cyclical breathing patterns, ranging from slow and calming to rapid and stimulating. It is recommended for relaxation, stress management, control of psycho physiological states and to improve organ function. In this pilot study Investigator recruited 24 type 2 diabetic patient and those who consent were provided with 6 days yoga course for a duration of 3 hours and trained to practice SKY at home for 12 week. At baseline and after 6 days of SKY, questionnaire on anxiety, depression and quality of life were provided to them. Biochemical parameters were measured at baseline and after 12 weeks of yoga. Two follow up yoga session were provided to the participants. Primary outcome were pre to post intervention change in the mental health and quality of life.

ELIGIBILITY:
Inclusion criteria

1. Patients showing stress as per the stress indicators.
2. Patients of both gender of age 30 to 65 years on oral anti diabetic agents
3. Patient is able to perform yoga postures and breathing exercise.
4. Patient is able to consent for the study.
5. Patient should be able to understand English as that is the medium used.

Exclusion criteria

1. Bipolar disorder
2. Antidepressant drugs
3. Type 1 diabetes
4. Pregnancy
5. Any acute coronary symptoms in past 6 months
6. Artificial pace-maker
7. Previous (SKY) or any type of spiritual meditation practiced within 6 months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of life | at 12 week
  change in score of Questionnaires on anxiety at 12 week of yoga intervention

SECONDARY OUTCOMES:
Improvement in HbA1c | at12 week of intervention
  Change in HbA1c value at 12 week of yoga intervention
Improvement in BMI | at 12 week of intervention
  Change in BMI at 12 week of yoga intervention
Improvement in lipid profile | at 12 week of intervention
  Change in lipid levels at 12 week of yoga intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Shiju, Mpharm, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait